CLINICAL TRIAL: NCT02856919
Title: A Multicenter, Open-label Clinical Trial to Evaluate the Efficacy and Safety of Once Daily Mirvaso® Gel (5 mg/g Brimonidine Tartrate) in Patients With Chronic Persistent Vascular Facial Erythema.
Brief Title: A Multicenter, Open-label Clinical Trial to Evaluate the Efficacy and Safety of Once Daily Mirvaso® Gel in Patients With Chronic Persistent Vascular Facial Erythema.
Acronym: BR14004
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma Brasil Ltda. (Industry)
Collaborators: Eurotrials Brasil Consultores Cientificos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR.14.004
Record Dates: First submitted 2016-07-19; First posted 2016-08-05 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-08

CONDITIONS: Chronic Persistent Vascular Facial Erythema
MeSH Terms: interventions — Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mirvaso® gel (Other): Mirvaso® gel (5 mg/g brimonidine tartrate)
  Interventions: Drug: brimonidine tartrate

INTERVENTIONS:
Drug: brimonidine tartrate — Mirvaso® gel (5 mg/g brimonidine tartrate)

SUMMARY:
This study evaluates the efficacy of Mirvaso® in the treatment of chronic persistent vascular facial erythema, after 4 weeks of treatment, by the Clinician erythema assessment.

DETAILED DESCRIPTION:
This is a multicenter, open-label trial in research participants with chronic persistent vascular facial erythema. All eligible research participants will receive Mirvaso® gel once daily for 4 weeks, and then will be followed-up for another 2 weeks.

The study will include 4 clinical visits: before Day 1, on Day 1, Day 29 and Week 6.

Within 5 days before Day 1, the research participant will have a screening visit for confirmation of eligibility.

On Day 1 and on Day 29, the research participant will have Mirvaso® gel applied, at the research site, and the evaluation will be conducted before application and 3 hours after application; During Days 2-28, research participants will have Mirvaso® gel applied once daily, at home; On Week 6, the research participants will go back to the research site for evaluation. No Mirvaso® gel will be applied after the visit on Day 29; Unscheduled visits may be performed during the trial for any safety reason.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female research participants aged 18 or higher.
2. Patients with chronic persistent facial erythema (at least 1 month before baseline [Day 1 hour 0]) of rosacea (with no restrictions to subtypes of rosacea), or originated from other dermatological condition, including, but not limited to seborrhoeic dermatitis, ulerythema ophryogenes, keratosis pillaris, microneedling, fractional radiofrequency, post-peeling treatments (medium depth and deep) or post-laser (ablative laser). Diagnosis is based on the investigator clinical judgement.
3. Clinician Erythema Assessment scores 2 (mild), 3 (moderate), or 4 (severe) at Day 1 prior to study treatment administration.
4. Patient Self-Evaluation scores 2 (mild), 3 (moderate), or 4 (severe) at Day 1 prior to study treatment administration.
5. Female patients with childbearing potential and negative pregnancy test at baseline. These patients should use a highly efficient contraceptive method during the study: combined oral contraceptives (estrogen and progesterone) or implanted contraceptives, or injectable contraceptives (with a stable dose for at least 1 month before study enrolment), bilateral tube ligation, hormonal intrauterine device (inserted at least 1 month before study entry), strict abstinence (at least 1 month prior to study entry and agreement in continuing throughout the study), or vasectomized partner (at least 3 months prior to study entry).
6. Female patients without childbearing potential (e.g., before menstruating, post-menopausal [absence of menstrual bleeding for 1 year prior to study entry], hysterectomy, or bilateral oophorectomy, less than one year after menopause).
7. Patients willing and able to fulfill the protocol requirements and duration.
8. Patients who understand and sign the Informed Consent Form at study inclusion, before any study procedure is carried out.

Exclusion Criteria:

- Any research participant that meets one or more of the following criteria is not eligible for the trial:

1. Female patients who are pregnant, breastfeeding or planning for pregnancy.
2. Current treatment with monoamine oxidase inhibitors, barbiturates, opiates, sedatives, systemic anesthetics or alpha agonists.
3. Patients who started or changed their doses of tricyclic antidepressants, cardiac glycosides, beta-blockers or other anti-hypertensive agents, in the 3 months prior to study entry.
4. Current diagnosis of Raynaud syndrome, thromboangiitis obliterans, orthostatic hypotension, severe cardiovascular disease, coronary or cerebral insufficiency, hepatic or renal failure, sclerodermia, Sjögren syndrome, or depression.
5. Any chronic or severe uncontrolled disease or medical chronic which may interfere with the interpretation of the study results, or may present a significant healthcare risk to the patient, if he/she participates in the study in accordance with the investigator judgment. (e.g. endocrine tumors, chromocytomas, systemic diseases that cause vascular erythema).
6. Known or suspected allergies or hypersensitivities to any of the components of the study treatments, including the active substance of brimonidine tartrate (see summary of product characteristics).
7. Patients who received, applied or ingested the following treatments in accordance with the time period specified before Day 1:

   * Topic facial treatments or procedures:

   Any dermatological/surgical facial procedure - 4 weeks. Immunomodulators (e.g. Methotrexate, Cyclosporin) - 4 weeks. Mirvaso® - 4 weeks.
   * Systemic treatments:

   Isotretinoin - 6 months. Immunomodulators - 90 days. Phototherapy - 4 weeks.
8. Exposure to excessive ultraviolet radiation within a week before Day 1 visit.
9. Presence of beard or excessive facial hair at Day 1, which interferes with the study treatment or study assessments and refusal to remove it during the study period.
10. Patients who do not wish to abstain from the use of forbidden medication or excessive exposure to ultraviolet radiation during the study period.
11. Vulnerable research participants (as deprived of freedom), in accordance with Section 1.61 of the International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use - ICH for Good Clinical Practices.
12. Current participation in any other clinical study with a drug or device OR participation within 30 days prior to Day 1 OR in an exclusion period of a previous clinical study (when possible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoints: Percentage of research participants with at least 1 degree of improvement from baseline in PSE on each moment of post-baseline evaluation | 1 year
  • Facial Erythema based on the Patient self-Evaluation (PSE) evaluated by the research participant on Day 1 (Hour 0 and Hour 3), Day 29 (Hour 0 and Hour 3). All eligible research participants will receive Mirvaso® gel once daily for 4 weeks.
  The study will include 4 clinical visits: before Day 1, on Day 1, Day 29 and Week 6.
  * Within 5 days before Day 1, the research participant will have a screening visit for confirmation of eligibility.
  * On Day 1 and on Day 29, the research participant will have Mirvaso® gel applied, at the research site, and the evaluation will be conducted before application and 3 hours after application;
  * During Days 2-28, research participants will have Mirvaso® gel applied once daily, at home;
  No Mirvaso® gel will be applied after the visit on Day 29;
  • Unscheduled visits may be performed during the trial for any safety reason.
Percentage of research participants with at least 1 degree of improvement from baseline in CEA on each moment of post-baseline evaluation. | 1 year
  • Facial Erythema based on the Clinician erythema assessment (CEA) evaluated by the investigator on Day 1 (Hour 0 and Hour 3), Day 29 (Hour 0 and Hour 3) . Clinician Erythema Assessment scores: 2 (mild), 3 (moderate), or 4 (severe) . All eligible research participants will receive Mirvaso® gel once daily for 4 weeks.
  The study will include 4 clinical visits: before Day 1, on Day 1, Day 29 and Week 6.
  * Within 5 days before Day 1, the research participant will have a screening visit for confirmation of eligibility.
  * On Day 1 and on Day 29, the research participant will have Mirvaso® gel applied, at the research site, and the evaluation will be conducted before application and 3 hours after application;
  * During Days 2-28, research participants will have Mirvaso® gel applied once daily, at home; No Mirvaso® gel will be applied after the visit on Day 29;
  * Unscheduled visits may be performed during the trial for any safety reason.

SECONDARY OUTCOMES:
Evaluate the efficacy of Mirvaso by the Patient Self Evaluation - PSE | 1 year
  To evaluate the efficacy of Mirvaso in the treatment of chronic persistent vascular facial erythema, after 4 and 6 weeks of treatment, by the patient self evaluation
Evaluate the efficacy of Mirvaso by the clinician erythema assessment - CEA | 1 year
  To evaluate the efficacy of Mirvaso in the treatment of chronic persistent vascular facial erythema, after 6 weeks of treatment, by the clinician erythema assessment.
Incidence of AEs. Evaluate the safety of Mirvaso | 1 year
  To evaluate the safety of Mirvaso up to 6 weeks after beginning the treatment
Study Participant Satisfaction Questionnaire | 1 year
  Research participants will fill the Study Participant Satisfaction Questionnaire at Hour 3 on Day 29 with 7 questions.
To evaluate the impact in the quality of life after 4 weeks of treatment with Mirvaso | 1 year
  Variation in the overall score in DLQI from baseline visit to each moment of post-baseline evaluation Dermatology life quality Index (DLQI) Questionnaire on Hour 0 on Day 1 and on Hour 3 on Day 29. 10 questions to measure how much the skin problem affected the quality life.
Variation in the overall score in FRQ from baseline visit to each moment of post-baseline evaluation | 1 year
  Variation in the overall score in FRQ from baseline visit to each moment of post-baseline evaluation Facial Redness Questionnaire (FRQ) on Hour 0 on Day 1 and on Hour 3 on Day 29. 12 questions to evaluate how much facial erythema (redness) is affecting life at the moment of answer.

OTHER OUTCOMES:
Instrumental Evaluation by Mexameter® | 1 year
  Evaluation by Mexameter®, including Day 1 (Hour 0 and Hour 3), Day 29 (Hour 0 and Hour 3) and Week 6. The equipment measures the main components of skin color, melanin and hemoglobin (erythema). This evaluation will only be performed in research sites where the necessary equipment is available.

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Instituto de Dermatologia e Estética do Brasil Ltda, Rio de Janeiro, Rio de Janeiro
  - Centro Brasileiro de Estudos em Dermatologia, Porto Alegre - RS, Rio Grande do Sul
  - Clinica Drmatologica Dra. Laura Buratini Ltda., Botucatu, São Paulo
  - Hosptial do Servidor Publico Municipal, São Paulo, São Paulo
  - Fundação do ABC, São Paulo, São Paulo